CLINICAL TRIAL: NCT06985472
Title: Orelabrutinib Combined With Zuberitamab in the Initial Treatment of MZL Single-arm, Multicenter Phase II Clinical Study
Brief Title: Orelabrutinib Combined With Zuberitamab in the Initial Treatment of MZL
Acronym: ZOOM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Zhiming (Other)
Responsible Party: Sponsor-Investigator, Li Zhiming, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-548-01
Record Dates: First submitted 2024-11-13; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Initial MZL; Untreated MZL; BTKi; CD20
Keywords: Orelabrutinib combined with Zuberitamab in the initial treatment of MZL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trial group (Experimental): Orelabrutinib combined with Zuberitamab for 6 cycles induction therapy, after that patients were treated with Orelabrutinib combined with Zuberitamab (administered every 2 cycles) for 6 cycles or had disease progression or toxicity intolerance.
  Interventions: Drug: ZO

INTERVENTIONS:
Drug: ZO — Orelabrutinib 150mg, po, gd, D1-D28, every 28 days, cycle 1-12; Zuberitamab: intravenously administered on day 1 of the cycle at a dose of 375mg/m2 every 28 days, once every cycle for cycles 1-6 and once every 2 cycles for cycles 7-12.

SUMMARY:
This is a multi-center, prospective cohort study. The main purpose of study is to evaluate the efficacy and safety of Orelabrutinib combined with Zuberitamab in the initial treatment of MZL Main efficacy indicators Complete response rate (CR) at the end of combination therapy.

DETAILED DESCRIPTION:
Marginal Zone Lymphoma (MZL) is a group of B-cell malignancies believed to originate from B lymphocytes, typically found in the marginal zones of lymphoid follicles in the spleen, lymph nodes, and mucosa-associated lymphoid tissues. Exploring more effective, low-toxicity treatment plans for MZL patients is a scientifically valuable and clinically significant attempt. With the development of new drugs, new drug regimens have become prominent in the treatment of MZL, and there is an increasing amount of research data on BTK inhibitors in the field of MZL. The BTK inhibitor Orelabrutinib has shown good efficacy in MZL and has been approved by the NMPA for the treatment of MZL in patients who have received at least one prior treatment.

This is a multi-center, prospective cohort study. The main purpose of study is to evaluate the efficacy and safety of Orelabrutinib combined with Zuberitamab in the initial treatment of MZL. After receiving 6 cycles of ZO regimen induction therapy, patients were treated with Orelabrutinib combined with Zuberitamab (administered every 2 cycles) for 6 cycles or had disease progression or toxicity intolerance. Main efficacy indicators Complete response rate (CR) at the end of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older; 2. ECOG performance status (PS) level 0~2; 3. The expected survival is not less than 12 weeks; 4. CD20-positive marginal area lymphoma confirmed according to WHO2008 lymphoma classification standard, including splenic MZL, lymph node MZL and extranodal MZL subtypes; 5. MZL with stage III/IV disease and stage I/II disease recurrence or progression after local treatment can also be included, and patients who have received BTKi inhibitor therapy for more than 6 months can also be included; 6. Enhanced computerized tomography/magnetic resonance imaging (CT/MRI) to detect measurable lesions; 7. Indications for MZL treatment that meet NCCN guidelines and have not received systematic treatment for MZL in the past (anti-infective treatment such as anti-HP and HCV is not systemic treatment); 8. The main organ function is normal and meet the following criteria :

1. blood routine examination standards must meet:

   1. ANC>1.0×109/L;
   2. PLT>75×109/L (≥50×109/L for patients with confirmed bone marrow infiltration);
   3. Hb>80g/dL;
2. Biochemical examination should meet the following criteria :

   1. TBIL<2×ULN;
   2. ALT and AST<2.5XULN(for patients with liver invasion,ALT and AST<5×ULN);
   3. Endogenous creatinine clearance ≥40ml/min (Cockcroft-Gault formula). 9. Women of childbearing age must have been using reliable contraception or had a pregnancy test (serum or urine) within 7 days of enrol with a negative result and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last dose of the test drug. For men, consent to use appropriate methods of contraception or surgical sterilization during the trial period and 8 weeks after the last dose of the trial drug; 10. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up.

      -

      Exclusion Criteria:
      1. Patients with central nervous system invasion;
      2. Previous or co-existing uncured malignancies, except cured skin basal cell MZL clinical trial protocol cancer, cervical carcinoma in situ and superficial bladder cancer;
      3. Patients with the following cardiovascular diseases: Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval 2450 ms for men and 2470 ms for women); According to NYHA standards, patients with grade III to V cardiac insufficiency or left ventricular ejection fraction (LVEF) <50% indicated by cardiac color ultrasound;
      4. Abnormal coagulation function (INR>1.5 or prothrombin time (PT) >ULN+4 seconds or APTT >1.5 ULN), have a tendency to hemorrhage or are receiving thrombolytic or anticoagulant therapy;
      5. Arteriovenous thrombosis events occurring in the 12 months prior to enrollment, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
      6. The presence of known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliac, coagulation disorder, thrombocytopenia, hypersplenism, etc.);
      7. Had major surgery or severe traumatic injury, fracture or ulcer within 4 weeks of enrollment;
      8. Have significant factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction;
      9. Active infections that require antimicrobial treatment (such as antimicrobial drugs, antiviral drugs, excluding chronic hepatitis B anti-hepatitis B treatment, antifungal drug treatment);
      10. Active hepatitis B (HBV DNA>2000IU/mL or 104 copy numbers /mL) or hepatitis C (hepatitis C antibody positive with HCVRNA higher than the lower detection limit of analytical methods);
      11. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
      12. Had participated in other anti-tumor drug clinical trials within 4 weeks before enrollment;
      13. Patients who had received potent CYP3A4 inhibitors within 7 days before enrollment, or had received potent CYP3A4 inducers within 12MZL clinical trial regimen days before enrollment;
      14. Pregnant or lactating women; A fertile patient who is unwilling or unable to take effective contraceptive measures;
      15. The investigator determines other circumstances that may affect the conduct of the clinical study and the determination of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1Y CRR | 2 years
  Complete response rate (CR) at the end of combination therapy Efficacy evaluation was performed every 3 cycles (12 weeks) during the treatment period, every 3 months during the maintenance treatment period, and every 3-6 months during the observation and follow-up period, using Lugano 2014 efficacy evaluation criteria. MRD tests are performed every 6 cycles within 2 years of starting the drug.For the main efficacy indicators, complete response rate (CR) and 95%CI were calculated.

SECONDARY OUTCOMES:
uMRD | 2 years
  Undetectable rate of total minimal residual lesions
  For the secondary efficacy indicators, such as 24-month progression-free survival (DFS) and 24-month overall survival (GFS), kaplan-Meier method was used to estimate and 95%CI were calculated, and survival curves were drawn. For secondary efficacy measures, uMRD, ORR and 95%CI were calculated.
ORR | 2 years
  Objective response rate
PFSR in 24m | 2 years
  24-month progression-free survival
OSR in 24m | 2 years
  24-month overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China